CLINICAL TRIAL: NCT03915418
Title: Validation of a Simple Method of Screening for Sleep Disorders in Children With Cerebral Palsy, Using Connected Tools
Brief Title: Validation of a Method of Screening for Sleep Disorders in Children With Cerebral Palsy, Using Connected Tools
Acronym: SOUTIEN-PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SOUTIEN-PC (29BRC18.0178)
Record Dates: First submitted 2018-12-07; First posted 2019-04-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Sleep Disorders
Keywords: Screening; sleep disorders; children; cerebral palsy; connected tools
MeSH Terms: conditions — Sleep Wake Disorders; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connected tools (Experimental): 1 night at home with connected tools only and 1 night at hospital with connected tools and PSG.
  Interventions: Procedure: Connected tools

INTERVENTIONS:
Procedure: Connected tools — At home, parents will record their child's sleep for 1night Then, on the date scheduled for the inclusion of the children and after the recording of the 1 night at home, the child will spend a night in a hospital environment to carry out the recording by polysomnography and tools connected simultaneously.

SUMMARY:
Cerebral palsy (CP) is the most common cause of child disability. Nearly 40% of PC children suffer from sleep disorders, which are not routinely screened. The neuro-cognitive, physical and environmental morbidity of sleep disorders should require their diagnosis and management. Limited access to the reference exam (polysomnography or PSG) delays the diagnosis and only allows screening of these disorders for a limited number of PC children. The hypothesis of our study is that connected technologies could optimize screening for sleep disorders in PC children by selecting children requiring PSG exploration and specific management.

ELIGIBILITY:
Inclusion Criteria:

* Boy or girl between 6 and 15 years old
* Confirmed diagnosis of cerebral palsy
* GMFCS class> 3
* Parents and child agreement

Exclusion Criteria:

* Pharmacological treatment of sleep disorders
* Diurnal and / or nocturnal ventilatory support
* Difficulty understanding and / or participation
* Subjects under 6 and over 15
* Refusal to participate
* Not affiliated with and not a beneficiary of a health insurance plan

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the diagnosis of sleep disorder | 15 days
  Sensitivity of sleep disorder diagnosis (positive / negative) obtained using connected tools in reference to that obtained by PSG
Specificity of the diagnosis of sleep disorder | 15 days
  Specificity of sleep disorder diagnosis (positive / negative) obtained using connected tools in reference to that obtained by PSG

SECONDARY OUTCOMES:
Diagnosis | 15 days
  Sensitivity and specificity of sleep disorder diagnosis using tools connected during 1 night at home (in comparaison with sleep disorder diagnosis using PSG)
Acceptability assessed by acceptability score for parents, and if possible children | 15 days
  Acceptability assessed by the acceptability score for parents, and if possible children, obtained by the SUS "System Usability Scale" scale. This questionnaire consists of ten questions to collect the subjective point of view of the user on the systems used
Sleep Quality Questionnaire | 15 days
  Sleep quality questionnaire used as a screening tool for sleep disorders: use of the Sleep Disturbance Scale for Children. Sleep Disturbance Scale for Children (SDSC) is a screening tool for sleep disorders in children and adolescents with good psychometric properties. It is one of the most used sleep questionnaires in the clinic but also in clinical research. Since its creation, the SDSC has been translated into several languages and recently validated in French. The ranking is obtained from a 26-item questionnaire completed by the parents. This scale distinguishes 6 major groups of sleep disorders: disorders of the installation or maintenance of sleep, breathing disorders, waking disorders, sleep-wake transition disorders, excessive daytime sleepiness and hypersudation of sleep.
Data quality outcome measures | 25 months
  Data quality will be assessed by establishing for each sensor the ratio (expressed in percent value) between the duration of the data effectively recorded to the total duration the patient weared the sensors. Pauses in recording during recording sessions will be identified in absolute value and duration for each sensor. Specific issues in recording will be reported, especially regarding the contents of RAW files.
A cost analysis of the sensor screening strategy will be compared to the PSG and the quality of life | 25 months
  A cost analysis of the sensor screening strategy will be compared to the PSG and the quality of life, measured as quality-adjusted life year QALY, will be simulated for one-year health conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Ropars, MD, Principal Investigator — Brest University Hospital in France
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - Fondation Ildys Ty-Yann, Brest
  - ESEAN Nantes, Nantes
  - AP-HP Hôpital Trousseau, Paris
  - Kerpape, Ploemeur